CLINICAL TRIAL: NCT02955771
Title: Multi-center, Randomized, Controlled, Open-label Study of Deuteporfin Photodynamic Therapy Plus Stenting Versus Stenting Alone as Treatment for Unresectable Advanced Perihilar Cholangiocarcinoma
Brief Title: Efficacy and Safety Study of PDT Using Deuteporfin for Unresectable Advanced Perihilar Cholangiocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDZJDTBF-NCC201512
Record Dates: First submitted 2016-11-02; First posted 2016-11-04 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Hilar Cholangiocarcinoma
Keywords: photodynamic therapy(PDT); stenting; Hilar Cholangiocarcinoma; Deuteporfin
MeSH Terms: conditions — Klatskin Tumor | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PDT-Deuteporfin（6 hour）plus stenting (Experimental): Deuteporfin (7.5mg/kg) was injected intravenously 6 hours before intraluminal photoactivation (wavelength,630 nm;light dose, 180 J/cm(2)). After PDT, endoscopic or percutaneous stenting will be performed.The second treatment may be given after 3 months.
  Interventions: Combination Product: PDT-Deuteporfin（6 hour); Device: stenting
- PDT-Deuteporfin（9 hour）plus stenting (Experimental): Deuteporfin (7.5mg/kg) was injected intravenously 9 hours before intraluminal photoactivation (wavelength,630 nm;light dose, 180 J/cm(2)). After PDT, endoscopic or percutaneous stenting will be performed.The second treatment may be given after 3 months.
  Interventions: Combination Product: PDT-Deuteporfin（9 hour); Device: stenting
- Stenting (Other): Endoscopic or percutaneous stenting alone will be performed.
  Interventions: Device: stenting

INTERVENTIONS:
Combination Product: PDT-Deuteporfin（6 hour) — Photodynamic therapy (PDT) involves the i.v. injection of Deuteporfin (7.5 mg/kg，Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd，Shanghai，China） followed by the illumination of the tumor. 6 hours after the injection,a laser light ( (wavelength,630 nm; light dose, 180 J/cm(2)；Guilin Xingda Photoelectric Medical Calinstrument Co., Ltd，,Fujian, China） will be applied to the tumor.The second courses of PDT may be given at 3-month intervals.
  Arms: PDT-Deuteporfin（6 hour）plus stenting
Combination Product: PDT-Deuteporfin（9 hour) — Photodynamic therapy (PDT) involves the i.v. injection of Deuteporfin (7.5 mg/kg，Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd，Shanghai，China) followed by the illumination of the tumor.9 hours after the injection,a laser light ( (wavelength,630 nm; light dose, 180 J/cm(2)；Guilin Xingda Photoelectric Medical Calinstrument Co., Ltd，,Fujian, China) will be applied to the tumor. The second courses of PDT may be given at 3-month intervals.
  Arms: PDT-Deuteporfin（9 hour）plus stenting
Device: stenting — The stenting procedure consists in the placement of plastic stents （Boston Scientific Corporation, MA,USA；or Cook Medical, Bloomington,USA）above the main tumors of the right and left hepatic bile ducts via endoscopic retrograde cholangiopancreatography (ERCP) or percutaneous transhepatic cholangiography (PTC).

SUMMARY:
This is a multi-center, randomized, controlled, open-label, phase IIa clinical study.The study will observe the efficacy and safety of Deuteporfin photodynamic therapy in addition to stenting compared to stenting alone in patients with unresectable advanced Perihilar Cholangiocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 18 or older.
* Diagnosed with radiologically and biopsy or cytology confirmed inoperable perihilar cholangiocarcinoma Bismuth Tumor Stage Ⅲ/Ⅳ.
* KPS≥70.
* Total Bilirubin<85.5 umol/L.
* Informed consent obtained.

Exclusion Criteria:

* The first diagnosis time of cholangiocarcinoma > 3 months before randomization.
* Expected survival <3 months.
* Patients with abnormal laboratory parameters: white blood cell<3.0×10(9)/L；hemoglobin <80g/L；Neutrophil Differential Count<1.5×10(9)/L；blood platelets<75×10(9)/L；or patients have other diseases of the blood system.
* Creatinine clearance >1.5×upper limit of normal range.
* Patients with severe liver function damage，or aspartate transaminase (AST) and/or alanine transaminase (ALT) >5×upper limit of normal range.
* Patients have intrahepatic metastasis, or distant metastasis (including distant lymph node metastasis); or bile duct cancer patients with other parts of the primary malignant tumor.
* Patients have activities of viral hepatitis, liver cirrhosis, liver abscess, alcoholic fatty liver, primary hepatocellular carcinoma, and other liver diseases; or patients have immunoglobulin G4 (IgG4) sclerosing cholangitis, primary sclerosing cholangitis, autoimmune cholangitis, and other cholangitis.
* Malignancies other than cholangiocarcinoma within 5 years prior to randomization, except for adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer.
* Patients had received PDT treatment prior to randomization.
* Patients had received bile duct carcinoma resection prior to randomization.
* Patients had received chemotherapy, or brachytherapy，or radiotherapy prior to randomization.
* Patients had received metal stent treatment prior to randomization.
* Presence of infection (active, untreated infection and/or acute bacterial or fungal infection) other than the infection of the bile duct (cholangitis).
* Uncontrolled severe hypertension [sitting systolic blood pressure (SBP) >180 mmHg and/or sitting diastolic blood pressure (DBP) >110 mmHg after medication]; have severe complications of hypertension or diabetes.
* Presence of severe heart, lung and central nervous system diseases.
* Presence of mental illness, or mental disorders can not accurately describe their feelings, or not according to the doctor's advice to take medication.
* History of alcohol abuse, drug abuse in the past 1 years.
* Presence of allergic diseases，or known to have light skin allergies or porphyria, or known to allergic to study drug(porphyrin drugs) or other similar compounds, cephalosporin antibiotics, other types penicillin, β lactamase inhibitors.
* Patients need to use prohibited drugs in proposal during the first 2 weeks of screening, or during the trial period.
* Patients having been enrolled in other clinical trial within 3 months prior to this clinical trial.
* Pregnant, lactating women or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception.
* The researchers weren't allowed to participate in this study as subjects.
* Patients unsuitable for enrollment in the clinical trial according to investigators decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
Overallsurvival | Up to 12 months
  From the date of randomization until the date of death or the last date the subject was known to be alive

SECONDARY OUTCOMES:
1-year survival rate | Up to 12 months
  From the date of randomization until the date of death or the last date the subject was known to be alive
The change rate of Bile duct stricture | Up to 6 months
  The date at the phase of baseline，at the end of first month, third month and sixth month
The change rate of serum bilirubin | Up to 1 month
  The date at the phase of baseline，at the first week ，at the end of first month
The change rate of carbohydrate antigen 199(CA199) | Up to 6 months
  The date at the phase of baseline，at the end of first month, third month and sixth month
The change rate of Karnofsky Performance Scale(KPS) | Up to 12 months
  From the date of randomization until the date of death or the last date the subject was known to be alive
The change rate of European Organization for Research and Treatment of Cancer Quality Of Life Questionnaire C30 (EORTC QLQ-C30) | Up to 12 months
  From the date of randomization until the date of death or the last date the subject was known to be alive

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyu Yin, MD. PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (4):
- China (4):
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Shanghai Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided